CLINICAL TRIAL: NCT00077246
Title: An Open-Label, Phase I/II Trial Of ABI-007 (A CREMOPHOR® El-Free, Protein Stabilized, Nanoparticle Paclitaxel) Administered Weekly In Chemotherapy Naive Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: ABI-007 in Treating Patients With Chemotherapy-Naïve Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000350076; MSKCC-03111; ABI-CA015
Record Dates: First submitted 2004-02-10; First posted 2004-02-11 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2009-12

CONDITIONS: Lung Cancer
Keywords: stage IV non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Taxes

INTERVENTIONS:
Drug: paclitaxel albumin-stabilized nanoparticle formulation

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as ABI-007, work in different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase I/II trial is studying the side effects and best dose of ABI-007 and to see how well it works in treating patients with stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose and dose-limiting toxicity of paclitaxel (albumin-stabilized Nanoparticle formulation) (ABI-007) in patients with chemotherapy-naïve stage IV non-small cell lung cancer.
* Determine the antitumor activity of this drug in these patients.
* Determine the safety and tolerability of this drug in these patients.

Secondary

* Determine the time to disease progression in patients treated with this drug.
* Determine duration of response in patients treated with this drug.
* Determine survival of patients treated with this drug.

OUTLINE: This is an open-label, dose-escalation study.

* Phase I: Patients receive paclitaxel (albumin-stabilized Nanoparticle formulation) (ABI-007) IV on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of ABI-007 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive ABI-007 as above at the MTD (determined in phase I). Patients are followed monthly for 6 months and then every 3 months for 1.5 years.

PROJECTED ACCRUAL: A total of 64 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed stage IV non-small cell lung cancer

  * Evidence of inoperable local recurrence or metastasis

    * Bone metastases or other nonmeasurable disease may not be only evidence of metastasis
* Measurable disease documented radiographically
* No evidence of active brain metastases or leptomeningeal involvement

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1 OR
* Karnofsky 80-100%

Life expectancy

* More than 12 weeks

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL

Hepatic

* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Bilirubin normal
* Alkaline phosphatase ≤ 2.5 times ULN (unless due to bone metastases and there is no radiologic evidence of hepatic metastases)

Renal

* Creatinine ≤ 1.5 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception for 1 month before and during study participation
* No prior allergy or hypersensitivity to study drug
* No other concurrent active malignancy
* No pre-existing peripheral neuropathy grade 1 or greater
* No other concurrent clinically significant illness
* No concurrent serious medical risk factor involving any of the major organ systems that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for metastatic disease
* More than 4 weeks since prior cytotoxic chemotherapy
* No concurrent doxorubicin
* No other concurrent taxanes
* No concurrent anthracyclines

Endocrine therapy

* Not specified

Radiotherapy

* At least 3 weeks since prior radiotherapy to a major bone marrow-containing area
* More than 4 weeks since prior radiotherapy except to a non-target lesion

  * Prior radiotherapy to a target lesion allowed provided there has been clear progression of the lesion since completion of radiotherapy

Surgery

* Not specified

Other

* Prior epidermal growth factor-targeted therapy allowed
* More than 4 weeks since prior investigational drugs
* No concurrent enrollment in another clinical trial in which investigational drugs are administered or investigational procedures are performed
* No concurrent treatment with any of the following:

  * Ritonavir
  * Saquinavir
  * Indinavir
  * Nelfinavir
* No concurrent anticonvulsants
* No other concurrent anticancer drugs
* No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2003-09; Primary Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) and dose-limiting toxicity (DLT) of ABI-007
Objective target lesion response (complete or partial) as measured by RECIST criteria

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events and serious adverse events
Nadir of myelosuppression
Changes in hematologic and clinical chemistry values
Changes in physical examination
Incidence of dose modifications, dose interruptions, and/or premature discontinuation of study treatment
Percentage of patients with stable disease for ≥ 16 weeks
Percentage of patients with complete or partial target response (total response)
Time to disease progression
Duration of response
Survival

CONTACTS AND LOCATIONS:
Overall Officials: Naiyer Rizvi, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Paik PK, James LP, Riely GJ, Azzoli CG, Miller VA, Ng KK, Sima CS, Heelan RT, Kris MG, Moore E, Rizvi NA. A phase 2 study of weekly albumin-bound paclitaxel (Abraxane(R)) given as a two-hour infusion. Cancer Chemother Pharmacol. 2011 Nov;68(5):1331-7. doi: 10.1007/s00280-011-1621-0. Epub 2011 Apr 3. PMID 21461889
- [Result] Rizvi NA, Riely GJ, Azzoli CG, Miller VA, Ng KK, Fiore J, Chia G, Brower M, Heelan R, Hawkins MJ, Kris MG. Phase I/II trial of weekly intravenous 130-nm albumin-bound paclitaxel as initial chemotherapy in patients with stage IV non-small-cell lung cancer. J Clin Oncol. 2008 Feb 1;26(4):639-43. doi: 10.1200/JCO.2007.10.8605. PMID 18235124